CLINICAL TRIAL: NCT06129721
Title: Emergent Stenting In Acute Vertebrobasilar Occlusions
Acronym: ESVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho Stroke International Services Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cuong Tran Chi, Director, Can Tho Stroke International Services Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESVO Study
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Acute Stroke; Ischemic Stroke, Acute; Vertebro Basilar Ischemia
Keywords: vertebrobasilar occlusions; acute ischemic stroke; emerging stenting
MeSH Terms: conditions — Stroke; Ischemic Stroke; Vertebrobasilar Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergent Stenting (Experimental): Emergent Stenting In Acute Vertebrobasilar Occlusions
  Interventions: Procedure: Emergent Stenting

INTERVENTIONS:
Procedure: Emergent Stenting — Emergent Stenting In Acute Vertebrobasilar Occlusions
  Other Names: ES

SUMMARY:
In the acute posterior circulation strokes, the vertebrobasilar occlusions frequently related to worse outcomes than the anterior ones. However, few studies mentioned the benefit and safety of the emergent stenting in the successful recanalization at these complex occlusions. The investigators investigated whether the improvement of clinical outcome was achieved in postprocedural 3-month.

DETAILED DESCRIPTION:
Acute ischemic stroke in posterior circulation account for nearly 20 - 25%, in which large vessel occlusions (LVOs) occur 0.8% - 5.7%. Although mechanical thrombectomy (MT) has recently been the gold standard in LVOs treatment, the futile recanalization (defined as unfavorable outcome despite early successful recanalization of target artery) rate was showed in posterior circulation higher than in anterior one. Multiple randomized controlled trials (BEST, BASICS, BAOCHE, ATTENTION) have recently reported the benefit of endovascular treatment better than of standard medical treatment for acute vertebrobasilar occlusions stroke. Besides, up to 36% LVOs with underlying intracranial stenosis and 64% with tandem lesions occured in the acute vertebrobasilar stroke. This was a reason why emergent stenting was considered to support the successful recanalization in the setting of failure of mechanical thrombectomy. Moreover, the successful recanalization is one of the independent predictors of good outcomes. However, the use of the loading dose dual antiplatelet therapy and peri-procedural complications made the safety of emergent stenting remain uncertain. Therefore, we aimed to investigate whether the impact of emergent stenting on the improved clinical outcome in vertebrobasilar occlusions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Onset to treatment time < 24 hours
* NIHSS ≥ 10
* pc-ASPECTS ≥ 5 on MRI

Exclusion Criteria:

* Premorbid mRS > 2
* Extensive, bilateral brain-stem infarction on neuroimaging
* Cerebellar mass effect on neuroimaging

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
The favorable 3-month outcome rate | 3 months
  The favorable 3-month outcome rate was accessed by modified Rankin Score (mRS), which comprised of included good (mRS 0 - ≤ 2) and fair (mRS 3).

SECONDARY OUTCOMES:
The symptomatic intracerebral hemorrhage rate | 24 hours after emergent stenting
  The symptomatic intracerebral hemorrhage was defined as patient's intracerebral hemorrhage with postprocedural mRS ≥ 5 and there were no other evident causes for the increased mRS

CONTACTS AND LOCATIONS:
Overall Officials: Cuong Tran Chi, Doctor, Study Director — Can Tho Stroke International Services General Hospital
Locations (1):
- Can Tho Stroke International Services Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tran CC, Le MT, Baxter BW, Nguyen-Luu G, Ngo MT, Nguyen-Dao NH, Duong-Hoang L, Mai-Van M, Nguyen MD. Rescue intracranial stenting in acute ischemic stroke: a preliminary Vietnamese study. Eur Rev Med Pharmacol Sci. 2022 Oct;26(19):6944-6952. doi: 10.26355/eurrev_202210_29875. PMID 36263574
- [Background] Le MT, Tran CC, Nguyen-Luu G, Ngo MT, Nguyen-Dao NH, Duong-Hoang L, Mai-Van M, Nguyen MD. Rescue stenting after the failure of intravenous thrombolysis and bridging thrombolysis: an initial Vietnamese report. Eur Rev Med Pharmacol Sci. 2022 Dec;26(24):9162-9169. doi: 10.26355/eurrev_202212_30667. PMID 36591828